CLINICAL TRIAL: NCT01740336
Title: A Phase II, Randomized Study of Paclitaxel With GDC-0941 Versus Paclitaxel With Placebo in Patients With Locally Recurrent or Metastatic Breast Cancer
Brief Title: A Study of Paclitaxel With GDC-0941 Versus Paclitaxel With Placebo in Participants With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO28509; 2012-003262-41 (EudraCT Number)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; Paclitaxel

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- A: Paclitaxel, GDC-0941 (Experimental): Participants will receive GDC-091 260 milligrams (mg) orally in repeated rounds of once daily (QD) dosing for 5 consecutive days followed by 2 consecutive days during which GDC-0941 will not be administered (5/7-day schedule). This 5/7-day schedule will be repeated weekly in each 28-day cycle until disease progression or intolerable toxicity. Participants will receive 90 milligrams per square meter (mg/m^2) intravenously (IV) weekly for 3 out of 4 weeks in every 28-day cycle.
  Interventions: Drug: GDC-0941; Drug: Paclitaxel
- B: Paclitaxel, Placebo (Placebo Comparator): Participants will receive placebo matching to GDC-0941 on the 5/7-day schedule along with 90 mg/m^2 IV weekly for 3 out of 4 weeks in every 28-day cycle.
  Interventions: Drug: Placebo; Drug: Paclitaxel

INTERVENTIONS:
Drug: GDC-0941 — GDC-0941 will be administered QD orally for 5 consecutive days each week.
  Arms: A: Paclitaxel, GDC-0941
Drug: Placebo — Placebo matching to GDC-0941
  Arms: B: Paclitaxel, Placebo
Drug: Paclitaxel — Paclitaxel will be administered IV weekly for 3 out of 4 weeks in every 28-day cycle.

SUMMARY:
This multicenter, randomized, single-blind, placebo-controlled, two arm study will evaluate the efficacy and safety of paclitaxel with GDC-0941 versus paclitaxel with placebo in participants with locally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast, with measurable or non-measurable locally recurrent or metastatic disease
* Human epidermal growth factor receptor 2 (HER2)-negative and hormone receptor (HR) (estrogen receptor and/or progesterone receptor)-positive disease as defined by local guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic and end organ function
* Women of childbearing potential must agree to remain abstinent or to use two adequate methods of contraception, including at least one method with a failure rate of less than (<) 1 percent (%) per year, during the treatment period and for at least 30 days after the last dose of study treatment or 6 months after discontinuation of paclitaxel, whichever is longer

Exclusion Criteria:

* Prior non-capecitabine chemotherapy for locally recurrent or metastatic disease
* Prior treatment with a phosphoinositide 3-kinase (PI3K) inhibitor for advanced or metastatic breast cancer
* History of intolerance to a taxane-containing therapy
* History of clinically significant cardiac or pulmonary dysfunction
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Clinically significant history of liver disease
* Active autoimmune disease or active inflammatory disease
* Immunocompromised status due to current known active infection with human immunodeficiency virus (HIV) or due to the use of immunosuppressive therapies for other conditions
* Need for current chronic corticosteroid therapy
* Pregnant, lactating, or breastfeeding women
* Current severe, uncontrolled systemic disease
* Known untreated or active central nervous system (CNS) metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2013-02-06 (Actual); Primary Completion 2015-10-20 (Actual); Study Completion 2015-12-10 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Assessed as per Modified Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) | From the time of randomization until disease progression or death from any cause (up to approximately 3 years)

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events | From randomization up to approximately 3 years
Percentage of Participants With Objective Tumor Response Assessed as per Modified RECIST v1.1 | From first observation of an objective tumor response until disease progression (up to approximately 3 years)
Percentage of Participants Acheiving Clinical Benefit (Partial Response, Complete Response or Stable Disease Lasting for at Least 6 Months) Assessed as per Modified RECIST v1.1 | From randomization until disease progression (up to approximately 3 years)
Duration of Confirmed Objective Response Assessed as per Modified RECIST v1.1 | From first observation of an objective tumor response until disease progression (up to approximately 3 years)
Population Pharmacokinetics (PK) for GDC-0941 | Day 8 of Cycle 1 and Day 1 of Cycle 6 (cycle length=28 days)
Population PK for Paclitaxel | Day 1 of Cycle 1 (cycle length=28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (97):
- United States (47):
  - Arizona Oncology Associates, PC - NAHOA, Sedona, Arizona
  - Pacific Cancer Medical Center, Anaheim, California
  - California Cancer Associates for Research & Excellence, Inc., Encinitas, California
  - Kaiser Permanente - Hayward, Hayward, California
  - Kaiser Permanente - Oakland, Oakland, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente - San Francisco (2238 Geary), San Francisco, California
  - University of California at San Francisco, San Francisco, California
  - Kaiser Permanente - San Jose, San Jose, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - Kaiser Permanente - South San Francisco, South San Francisco, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - Kaiser Permanente - Walnut Creek, Walnut Creek, California
  - Helen & Harry Gray Cancer Center-Hartford Hospital-CCD PRIME; Research, Hartford, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - Cancer Specialists of North Florida, Orange Park, Florida
  - Hematology - Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Joliet Oncology-Hematology; Associates, Ltd., Joliet, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Cotton-O'Neil Clinical Research Center, Hematology and Oncology; Cotton O'Neil Cancer Center, Topeka, Kansas
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Metairie Oncologist, LLC, Metairie, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Brookline, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Billings Clinic Cancer Center-CCD PRIME, Billings, Missouri
  - Nebraska Cancer Specialists; Oncology Hematology West, PC, Omaha, Nebraska
  - ProHEALTH Care Associates LLP, Lake Success, New York
  - Summa Health System, Akron, Ohio
  - Aultman Hospital; Aultman Hospital Cancer Center, Canton, Ohio
  - TriHealth Oncology Institute, Cincinnati, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Hematology and Oncology Associates of Sc, Greenville, South Carolina
  - Shivers Cancer Center at University Medical Center Brackenridge, Austin, Texas
  - Texas Oncology, Bedford, Texas
  - Texas Oncology, P.A. - El Paso; West, El Paso, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Texas Oncology, P.A. ;Sherman Cancer Center, Sherman, Texas
  - Northern Utah Associates, Ogden, Utah
  - Shenandoah Oncology Associates, Winchester, Virginia
  - Puget Sound Cancer Centers, Edmonds, Washington
  - Swedish Health Services, Seattle, Washington
- Australia (13):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Port Macquarie Base Hospital;North Coast Cancer Institute, Port Macquarie, New South Wales
  - Sydney Haematology & Oncology Clinic, Wahroonga, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Border Medical Oncology, Wodonga, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Adult Hospital, Mackay, Queensland
  - Ashford Cancer Center Research, Kurralta Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Bendigo Hospital; Oncology, Bendigo, Victoria
  - Peninsula and South Eastern Haematology and Oncology Grou, Frankston, Victoria
  - Royal Perth Hospital; Medical Oncology, Perth, Western Australia
- Austria (4):
  - Lkh-Univ. Klinikum Graz, Graz
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Krankenhaus Hietzing m.Neurolog. Zentrum Rosenhuegel, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - UZ Antwerpen, Edegem
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Ambroise Paré, Mons
  - Clinique Ste-Elisabeth, Namur
  - Sint Augustinus Wilrijk, Wilrijk
- Czechia (7):
  - Fakultni nemocnice Brno, Brno
  - Masarykuv onkologicky ustav, Brno
  - Krajska nemocnice Liberec a.s., Liberec
  - Multiscan s.r.o., Pardubice
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Nemocnice Na Bulovce, Prague
  - Thomayerova nemocnice, Praha 4 - Krc
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Institut Catala d´Oncologia Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital General Univ. Gregorio Maranon, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid
- United Kingdom (10):
  - Royal Sussex County Hospital, Brighton
  - Royal Surrey County Hospital, Guildford
  - Leicester Royal Infirmary, Leicester
  - Barts Hospital, London
  - The Christie, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals City Campus, Nottingham
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Royal Cornwall Hospital, Truro
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Vuylsteke P, Huizing M, Petrakova K, Roylance R, Laing R, Chan S, Abell F, Gendreau S, Rooney I, Apt D, Zhou J, Singel S, Fehrenbacher L. Pictilisib PI3Kinase inhibitor (a phosphatidylinositol 3-kinase [PI3K] inhibitor) plus paclitaxel for the treatment of hormone receptor-positive, HER2-negative, locally recurrent, or metastatic breast cancer: interim analysis of the multicentre, placebo-controlled, phase II randomised PEGGY study. Ann Oncol. 2016 Nov;27(11):2059-2066. doi: 10.1093/annonc/mdw320. Epub 2016 Aug 29. PMID 27573562